CLINICAL TRIAL: NCT05703243
Title: Discovering Novel Cancer Treatment Options Using a Comprehensive NGS-based Liquid Molecular Testing Panel in the Community Setting. ("DINOSAur II")
Brief Title: Discovering Novel Cancer Treatment Options Using a Comprehensive NGS-based Liquid Molecular Testing Panel in the Community Setting ("DINOSAur II")
Acronym: DINOSAur II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glendale Adventist Medical Center d/b/a Adventist Health Glendale (Other)
Collaborators: Guardant Health, Inc. (Industry)
Responsible Party: Principal Investigator, Mihran Shirinian, Principal Investigator, Glendale Adventist Medical Center d/b/a Adventist Health Glendale
Other Study IDs: DINOSAur II
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Stage III Solid Tumors; Stage IV Solid Tumors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active: Newly diagnosed cancer patients.
  Interventions: Diagnostic Test: Comprehensive liquid molecular panel test; Other: EORTC QLQ-30
- Control: Historically diagnosed cancer patients.

INTERVENTIONS:
Diagnostic Test: Comprehensive liquid molecular panel test — Lab test
  Groups: Active
Other: EORTC QLQ-30 — Quality of life questionnaire
  Groups: Active

SUMMARY:
To prospectively identify cancer patients whose tumors express specific molecular markers targeted by therapeutic agents from a comprehensive l i q u i d molecular test, for the purpose of selecting the most clinically appropriate treatment in a pragmatic two arm trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent in accordance with the methods and procedures of this study
* Diagnosis of cancer (stage 3 and stage 4; solid tumors only) requiring medical care
* Patients who have not received treatment related to his/her cancer
* Patients who are willing to sign a release of medical records to the research team
* Male and female patients ≥18 years of age
* Patients under oncology care
* Sufficient clinical status for collection of blood sample within usual care

Exclusion Criteria:

* Patients considered minors in the jurisdiction where the protocol is conducted
* Patients who are prisoners and pregnant women
* Patients who cannot provide consent and did not sign a power of attorney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed cancer patients at the pathology level
Sampling Method: Probability Sample
Enrollment: 572 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (QLQ-C30) | 2 years
  The EORTC Core Questionnaire (QLQ-C30) includes six clearly distinguishable functioning scales that have been thoroughly tested and validated on an international level and that are available in 110 different language versions. The scaling of items is 1 (Not at all) to 4 (Very much), 1 (Very poor) to 7 (Excellent). The higher the score the better the quality of life.

SECONDARY OUTCOMES:
Compare the proportion of enrolling in clinical trials | 2 years
  To compare the proportion of enrolling in clinical trials between cancers patients who received the CLMT versus cancer patients with no CLMT.

CONTACTS AND LOCATIONS:
Overall Officials: Mihran H Shirinian, MD, Principal Investigator — Glendale Adventist Medical Center dba Adventist Health Glendale
Locations (1):
- Adventist Health Glendale, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No